CLINICAL TRIAL: NCT05669547
Title: Dual Hormone Closed Loop in Type 1 Diabetes: a Randomized Trial (DARE)
Brief Title: Dual Hormone Closed Loop in Type 1 Diabetes
Acronym: DARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch National Health Care Institute (Other); Inreda Diabetic B.V. (Industry)
Responsible Party: Principal Investigator, Thomas van Sloten, Principal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22/671
Record Dates: First submitted 2022-11-22; First posted 2023-01-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes type1; Diabetes
Keywords: dual hormone; fully closed loop; bihormonal pump; artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients currently on multiple daily injections (MDI) + continuous or flash glucose monitoring (CGM; FGM) or on a hybrid closed loop (HCL).
- Intervention (Experimental): Patients on dual hormone fully closed loop (DHFCL) therapy.
  Interventions: Device: dual hormone fully closed loop (DHFCL)

INTERVENTIONS:
Device: dual hormone fully closed loop (DHFCL) — dual hormone fully closed loop consisting of an algorithm, sensors and both insulin and glucagon infusion.
  Other Names: Inreda AP (Inreda Diabetic BV)
  Arms: Intervention

SUMMARY:
This study is a 12 month open-label, two-arm randomised parallel-group trial in adult type 1 diabetes patients executed in 14 centres in the Netherlands. The aim of this study is to determine the long-term clinical effectiveness of treatment with a dual-hormone (insulin and glucagon) fully closed loop system during 12 months compared to the current most used care and to the currently most advanced technological care. Secondary objectives include the assessment of cost-effectiveness, Patient Reported Outcome Measures (PROMs), other glycaemic outcomes and safety.

DETAILED DESCRIPTION:
Rationale: Patients with type 1 diabetes mellitus (T1DM) require lifelong insulin therapy. Insulin therapy improves but does not fully normalise blood glucose levels with current therapies. Current therapies include subcutaneous insulin injection or subcutaneous insulin infusion, combined with a device to measure glucose levels (finger stick, intermittent sensor or continuous glucose monitoring). Although having provided a huge improvement in glycaemic control, patients have to work hard every day and still have to calculate mealtime boluses. An automated insulin delivery device covering both basal and prandial insulin requirement would mean another great leap forwards. The dual-hormone fully closed loop (DHFCL) provides such a new strategy of automated insulin delivery coupled with targeted glucagon infusion as insulin-antagonist to even more approximate normal physiology.

Objective: To determine the long-term clinical effectiveness of treatment with a dual-hormone (insulin and glucagon) fully closed loop system during 12 months compared to the current most used care and to the currently most advanced technological care. Secondary objectives include the assessment of cost-effectiveness, Patient Reported Outcome Measures (PROMs), other glycaemic outcomes and safety.

Study design: A 12 month open-label, two-arm randomised parallel-group trial. Study population: Adult (age ≥18 years) patients with T1DM for at least 1 year with an HbA1c at entry ≤ 91 mmol/mol.

Intervention: The study includes two separately randomised arms, defined by current diabetes treatment. In one arm, patients currently on Multiple Daily Injections (MDI; at least once daily long-acting insulin and thrice daily short-acting insulin) in combination with continuous or flash glucose monitoring (CGM or FGM; currently the most used strategy) are 1:1 randomised to either the intervention, i.e. the DHFCL, or continuation of their current treatment. In the other arm, patients currently on hybrid closed loop treatment (HCL; presently the most advanced diabetes control treatment) are 1:1 randomised to either the intervention or continuation of their current care.

Main study parameters/endpoints: The main study endpoint is the Time in Range (TIR; % of time spent in the 3.9-10 mmol/l target range) at 12 months, which will be compared between the intervention and the control treatment within each arm. Secondary endpoints include cost-effectiveness, PROMs, other glycaemic outcomes, safety measures and device-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years;
* Diagnosed with type 1 diabetes mellitus at least one year ago;
* HbA1c ≤ 91 mmol/mol;
* Treated with either MDI with FGM/CGM or treated with HCL:

  * MDI+FGM/CGM for ≥ 3 months with an adequate sensor use during at least 70% of the time in the month prior to screening (based on sensor usage from the download summary report of the FGM/CGM);
  * HCL for ≥ 3 months with a frequency of use ≥ 70% of the time in auto mode over the previous month prior to screening;
* Does not reach the treatment goals over the last 8 weeks:

  * for MDI+FGM/CGM: subject has a TIR <80% or Time Below Range (TBR) >4%;
  * for HCL: subject has a TIR <80% or TBR >4%;
* Willing to take or switch to insulin Humalog when randomized to the intervention DHFCL arm;
* Under treatment in one of the participating centres;
* Willing and able to sign informed consent;
* Access to internet at home (for DHFCL data upload).

Exclusion Criteria:

* Current use of non-approved HCL device;
* BMI >35 kg/m2;
* eGFR<30 mL/min/1.73m2;
* Plan to change usual diabetes regimen in the next 3 months;
* Current participation in another diabetes-related clinical trial;
* Actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or device in the last 2 weeks before enrolment into this study, as per investigator judgment;
* Established history of allergy or severe reaction to adhesive or tape that must be used in the study;
* Use of oral glucose-lowering medication;
* Active retinopathy or painful neuropathy;
* Daily use of acetaminophen during the trial (all arms), as this may influence the sensor glucose measurements. Incidental use with a maximum of e.g. 3 daily doses of 1000mg paracetamol for a maximum of 3 consecutive days is allowed
* Limited ability to see, and to hear or feel alarm signals of the closed loop system;
* Current pregnancy, breast feeding or planning to become pregnant in the 12 months of the trial or using ineffective birth control methods;
* Presence of a medical or psychiatric condition, longstanding serious adherence problems, anticipated problems in handing over diabetes control to a device or use of a medication that, in the judgment of the investigator, clinical protocol chair, or medical monitor, could compromise the results of the study or the safety of the participant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Time in Range (TIR) at 12 months (measured with an independent FSL Pro IQ sensor) | 12 months
  TIR (% of time spent in the 3.9-10 mmol/l target range) at 12 months, which will be compared between the intervention and the control treatment within each arm.

SECONDARY OUTCOMES:
World Health Organization-Five Well-Being Index (WHO-5) score (Patient reported outcomes (PROMs) | at 0, 3, 6, 9 and 12 months
  The World Health Organisation- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing.
Health-related quality of life scores (EQ-5D-5L) (Patient reported outcomes (PROMs) | at 0, 3, 6, 9 and 12 months
  As described on the Euroqol website, the EQ-5D-5L measures mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Problem Areas In Diabetes (PAID-5) score (Patient reported outcomes (PROMs) | at 0, 3, 6, 9 and 12 months
  Evaluates problem areas in diabetes
Diabetes Treatment and Satisfaction Questionnaire status and change (DTSQ-s and DTSQ-c) scores (Patient reported outcomes (PROMs) | at 0, 3, 6, 9 and 12 months
  Measurement of treatment satisfaction
Hypoglycaemia Fear Survey-II (HFS-II) Worry subscale score; (Patient reported outcomes (PROMs) | at 0, 3, 6, 9 and 12 months
  Measures hypoglycaemia fear
Pittsburgh Sleep Quality Index score (Patient reported outcomes (PROMs) | at 0, 3, 6, 9 and 12 months
  Measures sleep quality and duration
Insulin delivery systems: perceptions, ideas, reflections and expectations (INSPIRE) scores (Patient reported outcomes (PROMs) | at 0, 3, 6, 9 and 12 months
  Measures ideas, perceptions and expectations of the insulin device - only for HCL (control) and DHFCL groups
Hypoglycaemia unawareness (Gold-Clarke) (Patient reported outcomes (PROMs) | at 0 and 12 months
  Measurement of hypoglycaemia unawareness
Cost-effectiveness: cost per quality adjusted life year. | 12 months
  To determine the cost-effectiveness of treatment with the DHFCL. Including data:
  Medical Consumption Questionnaire (MCQ), at 0, 3, 6, 9 and 12 months; Productivity Cost Questionnaire (PCQ), at 0, 3, 6, 9 and 12 months; Detailed hospital health care consumption for each individual patient (collected from electronic patient files, including unplanned contact moments) Cost effectiveness: cost per quality adjusted life year.
Other glycaemic outcomes | at 0, 3, 6, 9 and 12 months
  Including Time Below Range (TBR), Time Above Range (TAR), glycaemic variability, number of hypoglycemic events and HbA1c.
Time Above Range (TAR) Other glycaemic outcomes | at 0, 3, 6, 9 and 12 months
  Measured with an independent Freestyle Libre Pro IQ sensor
  * level 1 and 2 hyperglycaemia: >10.0 mmol/l;
  * level 2 hyperglycaemia: >13.9 mmol/l;
Time Below Range (TBR) Other glycaemic outcomes | at 0, 3, 6, 9 and 12 months
  Measured with an independent Freestyle Libre Pro IQ sensor
  * level 1 and 2 hypoglycaemia: <3.9 mmol/l;
  * level 2 hypoglycaemia: <3.0 mmol/l;
Number of hypoglycaemic events Other glycaemic outcomes | at 0, 3, 6, 9 and 12 months
  Measured with an independent Freestyle Libre Pro IQ sensor defined as glucose <3.0 mmol/l for 15 consecutive minutes when the time between two successive events is less than 30 minutes, they will be combined and counted as one event
Mean glucose Other glycaemic outcomes | at 0, 3, 6, 9 and 12 months
  Measured with an independent Freestyle Libre Pro IQ sensor
  * day and night;
  * day: from 06:00 to 23:59 hours;
  * night: from 00:00 to 05:59 hours;
Glycaemic variability Other glycaemic outcomes | at 0, 3, 6, 9 and 12 months
  Based on independent Freestyle Libre Pro IQ sensor data
  * Coefficient of variation;
  * Standard deviation.
HbA1c Other glycaemic outcomes | at 0, 3, 6, 9 and 12 months
  venipuncture
  * Mean;
  * Percentage patients achieving HbA1c ≤ 53 mmol/mol.
Long-term safety outcomes | 12 months
  To assess long-term safety of the DHFCL, including the incidence of (severe) adverse events, incidence of device issues and the effects of excluding daily use of acetaminophen on non steroidal inflammatory drug (NSAIDs) use and associated drug complications rate.
Daily insulin use (units/day) DHFCL outcomes | at 3, 6, 9 and 12 months
  Measured by DHFCL device
daily glucagon use.DHFCL outcomes | at 3, 6, 9 and 12 months
  Measured by DHFCL device Daily insulin use, daily glucagon use and percentage of time glucose control algorithm active at 0, 3, 6, 9 and 12 months.
Percentage of time glucose control algorithm active DHFCL outcomes | at 3, 6, 9 and 12 months
  Measured by DHFCL device

OTHER OUTCOMES:
Patient reported daily insulin use control group | at 3, 6, 9 and 12 months
  The amount of daily insulin use reported by the patients in the control group
Weight (kg) at baseline and 12 months | 12 months
  Change of weight 0-12 months
Blood pressure (SBP/DBP in mmHg) at baseline and 12 months | 12 months
  Change of blood pressure and heart rate 0-12 months
Heart rate (/min) at baseline and 12 months | 12 months
  Change of heart rate 0-12 months
Frequency of unplanned patient contact with the diabetes team | at 3, 6, 9 and 12 months
  Evaluating whether the DHFCL imposes more unplanned patient contact moments
Concomitant medication, at screening, baseline, 3, 6, 9 and 12 months | at screening, baseline, 3, 6, 9 and 12 months
  Evaluation of medication
Continuation rate of the DHFCL | at 12 months
  Expressed as the percentage of participants that continue DHFCL treatment after 1 year of use
Reasons for discontinuation of the DHFCL treatment. | at 3, 6, 9 and 12 months
  Patients will be asked by the physician what the reason of discontinuation is when discontinuing the DHFCL treatment before the end of study

CONTACTS AND LOCATIONS:
Locations (14):
- Netherlands (14):
  - Meander MC, Amersfoort
  - Amsterdam UMC, AMC, Amsterdam
  - Amsterdam UMC, VUmc, Amsterdam
  - OLVG, Amsterdam
  - Gelre Ziekenhuis, Apeldoorn
  - Rijnstate, Arnhem
  - Catharina Ziekenhuis, Eindhoven
  - Martini Ziekenhuis, Groningen
  - UMC Groningen, Groningen
  - Tergooi Ziekenhuis, Hilversum
  - LUMC, Leiden
  - St. Antonius, Nieuwegein
  - UMC Utrecht, Utrecht
  - Isala Klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jancev M, Snoek FJ, Frederix GWJ, Knottnerus H, Blauw H, Witkop M, Moons KGM, van Bon AC, DeVries JH, Serne EH, van Sloten TT, de Valk HW; DARE study consortium. Dual hormone fully closed loop in type 1 diabetes: a randomised trial in the Netherlands - study protocol. BMJ Open. 2023 Aug 23;13(8):e074984. doi: 10.1136/bmjopen-2023-074984. PMID 37612114
- See also: DARE trial website (Dutch) — https://darestudie.nl

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT05669547/SAP_000.pdf